CLINICAL TRIAL: NCT03506230
Title: The Effect of Financial Incentives on Improvement of Glycemic Control in Diabetic Patients From Low Socioeconomic Background
Brief Title: Financial Incentives for Low Socioeconomic Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0159-15
Record Dates: First submitted 2018-03-25; First posted 2018-04-24 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Rewards; Medication Adherence; Health Behavior; Diabetes Mellitus; Copayments
MeSH Terms: conditions — Medication Adherence; Health Behavior; Diabetes Mellitus | interventions — Fertility

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the intervention group and the control group. The randomization will be in blocks of 6. In addition, the randomization will be in strata according to the level of HbA1c: 8.5% <HbA1c> 9.5%, 9.6%> HbA1c> 11%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentives group (Experimental): a bonus to buy their medications if they improve their HbA1c
  Interventions: Behavioral: Incentives
- Standard group (No Intervention): Will buy their medications as usual

INTERVENTIONS:
Behavioral: Incentives — A bonus to buy their medications if they reduce their HBA1c
  Arms: Incentives group

SUMMARY:
Patients with uncontrolled diabetes [glycated hemoglobin (Hba1c)>8.5%] from low socioeconomic status neighborhoods in Jerusalem will be recruited. They will be randomly assigned to an intervention group and a control group. The intervention group will be offered a bonus to buy their medications, 100 Israeli Shekels (ILS) (30$) each month for 3 months, if they reduce their HBA1c by 0.7% or if their HbA1c level reaches 7.5%. After 6 months they will be eligible for another bonus for one month if they improve their HbA1c by 0.3% from the previous test. The control group will buy medications as usual. All participants will be contacted by phone and will be encouraged to contact their doctor, to perform blood tests and to maintain a healthy lifestyle.

DETAILED DESCRIPTION:
The study will be performed in primary care clinics in a big Health Funds in Jerusalem and the area (Clalit Health Services). Guidance will be given to the professional staff in the clinics and the pharmacists in the pharmacies of the Health Care Fund. Candidates will be identified from lists of diabetic patients and will be invited to the clinic or will be contacted upon arrival to the clinic. Candidates that will agree to participate in the study will sign an informed consent and answer a small survey.

Candidates that do not have a recent HbA1c result (from the last month) will be referred to perform a blood test. Only patients with an updated result of 8.5% or higher, will be included in the study. The participants will receive explanations from the research staff or the medical professionals at the clinic. General recommendations for diabetes care will be provided orally, and a written summary will be given. Contact details with the research staff will be provided as well.

All participants will be contacted by phone to inform them of their group membership within three days of the recruitment, or 3 days after receiving the result of the blood test. The information will be delivered by a member of the research team that will not know the participants. The result will be sent by mail as well.

The incentives group participants will be told they will receive a bonus to buy their medications at the designated pharmacies. After three months, if they reduce their HBA1c by 0.7% compared to the previous test, or if their HbA1c level is reduced to 7.5% or below, they will get a bonus of up to 100 ILS (30$) every month, for the next three months depending on the total amount of their purchased medicine that month. Six months after entering the trial they will be entitled to a bonus for one additional month if they have reduced their HbA1c level by 0.3% compared to the last test. The bonus can be used to pay for chronic prescription drugs for diabetes, hypertension (HTN) or hyperlipidemia those who are included in the Israeli "health basket," or not included.

The standard treatment group will buy medications as usual. All participants will be encouraged to get their treatment and prescriptions from their physician, and to take their medication regularly. They will receive recommendations for a healthy lifestyle with low-sugar diet and physical activity, be encouraged to perform routine blood and urine tests and have an eye examination once a year. They will receive by mail a tracking page for documentation of hypoglycemia events. They will be asked to document events of symptomatic low blood sugar (55mg/dl or less) and to indicate whether they needed help to recover from hypoglycemia. They will be told a research assistant will contact them during the follow- up period.

The research assistant will call all participants at one, three, four and six months after the entrance to the study. The patients will be reminded to perform blood tests after three months and six months, to refer to their doctor to get their treatment and prescriptions, and to comply with all other recommendations mentioned above. These frequent calls will be performed to ensure patients safety.

The patients will be asked by phone about symptoms of hypoglycemia with sugar levels of 55 mg/dl or lower, loss of consciousness or need of intervention to increase their blood sugar, what kind of help was needed, and if they went or were taken to the hospital. Severe hypoglycemic events will be reported immediately to the research coordinator, to the attending physician and the ethics committee.

The procedure of the medications bonuses will be arranged in advance with the health maintenance organization (HMO) pharmacies. The patients will get vouchers for buying medications from their doctor or the research staff. Patients from the incentive group will be allowed to receive both bonuses (after three months and after six months) only if they perform their blood tests as scheduled. A patient that will delay his test to four months or more from entry will be entitled only to the first three months bonus. This result will count as the final result for this patient. At six months, participants of all groups will be encouraged to perform their blood tests.

At the end of the trial, data will be collected from the medical records, including HbA1c result, performance of LDL-Cholesterol, triglyceride (TG), albumin-creatinine ratio during the last year test and an eye examination during the last year, consultations with the attending doctor or the diabetic specialist that included prescribing medications for diabetes, name of the patient's clinic, co-morbidities (cardiovascular, respiratory, renal and vascular), diabetes complications, number of medications for diabetes, and prescription of newer medications for diabetes (Dipeptidyl peptidase-4 (DPP4) inhibitors, glucagon-like peptide glycolipoprotein (GLP) 1 agonists, Sodium-dependent glucose cotransporters (SGLT) 2 inhibitors). Information about hypoglycemia events will be drawn from the medical files as well: episodes of severe hypoglycemia, when the patient needed the help of another person, or capillary blood glucose testing of 55 mg/dl or below accompanied with symptoms, visits to the emergency room attributed to hypoglycemia, Finally, hospitalizations for a week or more, and regular discount for medications due to low income.

The recruitments stage will last one year. Each participant will take part in the study for 6 months, not more than 7 months, till they perform the last blood test. After the last participant performs the final blood test, there will be an ending period for 6 months. Altogether the study will be carried out for two years.

The sample size was estimated for the primary outcome, of 0.55% difference in HbA1c levels between the intervention and the control group, and a 1.2 standard deviation of HbA1c tests of diabetic patients in Clalit Health Services in 2013. In this study, the effect is expected to be higher as in low socioeconomic status patients. To ensure an 80% power to detect differences between arms, and a significance level of 0.05 (two-sided), 76 participants will be needed in each group. To account for dropouts 15% additional participants will be recruited, or a total number of 180 participants.

Any information of severe hypoglycemia will be immediately reported to a research team member to examine the event and to report to the attending physician and the chief investigator. In this situation, the patient's participation in the research will be discontinued, and the event will be reported to the Ethics Committee. In case of death for any reason, it will be reported in detail to the Ethics Committee. An interim analysis will be conducted after half of the study participants (84 people) will finish their study to test the safety of the study.

The researchers will allow visitors on behalf of the ethics committee or regulators to have direct access to information sources and other documents. Monitoring and auditing will take place after half of the participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes for at least 6 months
* Diabetes for a maximum of ten years
* Updated HbA1c level of between 8.5 and 11% from the last month
* Agreement to participate and sign an informed consent

Exclusion Criteria:

* Pregnancy
* Insulin therapy
* Psychiatric disorder from the first or second line according to the Diagnostic and Statistical Manual of mental disorders (DSM)
* Active oncology disease [excluding squamous cell carcinoma (SCC) and basal cell carcinoma (BCC)
* Planed bariatric surgery for the next 6 months
* Cardiac hospitalization in the previous year
* A severe hypoglycemia event three months prior to allocation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Differences in HbA1c after six months | Six months
  Differences between the groups in the change in HbA1c between the test at the entrance to the study and the test six months later

SECONDARY OUTCOMES:
Differences in HbA1c after three months | 3 months
  Differences between the groups in the change in HbA1c between the test at the entrance to the study and the test three months later
Differences in the proportion of participants who improved their HbA1c by 1% or more | Six months
  Differences between the groups in the proportion of participants who improved their HbA1c by 1% or more between the test at the entrance to the study and the test after six months
Whether or not HbA1c test was performed at 3 months | Two months
  Differences between groups in whether or not HbA1c test was performed at 3 months

OTHER OUTCOMES:
Whether LDL cholesterol test was performed | Six months
  Differences between the groups whether or not LDL cholesterol test was performed during the study period
Performing a urine microalbumin test | Six months
  Differences between the groups in performing or not a urine microalbumin testing
Differences in the number of GP visits | Six months
  Differences in the number of visits to a general practitioner (GP) according to the medical records in which prescriptions for diabetes medications were prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Lahad, MD, MPH, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit health services, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long JA, Jahnle EC, Richardson DM, Loewenstein G, Volpp KG. Peer mentoring and financial incentives to improve glucose control in African American veterans: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):416-24. doi: 10.7326/0003-4819-156-6-201203200-00004. PMID 22431674
- [Background] Tarasiuk A, Reznor G, Greenberg-Dotan S, Reuveni H. Financial incentive increases CPAP acceptance in patients from low socioeconomic background. PLoS One. 2012;7(3):e33178. doi: 10.1371/journal.pone.0033178. Epub 2012 Mar 30. PMID 22479368